CLINICAL TRIAL: NCT02524054
Title: Aerosol Inhalation Treatment for Dyspnea
Brief Title: Aerosol Inhalation Treatment for Dyspnea - Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Robert Banzett, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2011P000027; R01NR012009 (NIH)
Record Dates: First submitted 2015-05-05; First posted 2015-08-14 (Estimated); Results first posted 2017-10-13 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Dyspnea
Keywords: Dyspnea; Hospitalized patients; Ambulatory outpatients; Shortness of breath; Chronic obstructive pulmonary disease; Pulmonary disease
MeSH Terms: conditions — Dyspnea; Pulmonary Disease, Chronic Obstructive; Lung Diseases | interventions — Furosemide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aerosol furosemide Study 2a (Experimental): Subjects will inhale 40mg of furosemide aerosol over the course of 10-15 min. This will be a single, unblinded administration.
  Interventions: Drug: Furosemide
- Aerosol furosemide Study 2b Arm F (Experimental): Inhalation of furosemide aerosol one one day then placebo saline aerosol on another day. Baseline measurement 15 min; Inhalation over the course of 10-15 min.; outcome measurement 15 min. Watch for adverse effects 2 hours.
  Interventions: Drug: Furosemide; Drug: Aerosolized saline
- Aerosol furosemide Study 2b Arm S (Experimental): Inhalation of saline aerosol one one day then furosemide aerosol on another day. Baseline measurement 15 min; Inhalation over the course of 10-15 min.; outcome measurement 15 min. Watch for adverse effects 2 hours.
  Interventions: Drug: Furosemide; Drug: Aerosolized saline

INTERVENTIONS:
Drug: Furosemide — 80 mg of Furosemide in 8ml saline will be aerosolized using ultrasonic screen nebulizers. Aerosol will be delivered using a clinical volume-control ventilator to regulate inspiratory flow and volume.
  Other Names: Lasix
Drug: Aerosolized saline — 8ml saline will be aerosolized using ultrasonic screen nebulizers. Aerosol will be delivered using a clinical volume-control ventilator to regulate inspiratory flow and volume.
  Other Names: Placebo
  Arms: Aerosol furosemide Study 2b Arm F; Aerosol furosemide Study 2b Arm S

SUMMARY:
The purpose of this protocol is to develop and test aerosol furosemide, as a treatment that has the potential to significantly improve symptom management and enhance the quality of care for patients with intractable dyspnea.

DETAILED DESCRIPTION:
This is the second study in a series of studies investigating the treatment effect of aerosolized furosemide on hospitalized patients and outpatients with intractable dyspnea. The study will focus on patients who experience intractable dyspnea at rest or with minimal activity, e.g., dressing, bathing, cooking, or walking stairs or short distances.

There are two parts to this study: Study 2a is a pilot study on 5-10 patients. These trials are not blinded or placebo controlled; the investigators will use them to discover practical problems, and take the information back to the laboratory to develop solutions. We enrolled 7 subjects for Study 2a.

Study 2b will a randomized, placebo - controlled, double- blind study on 25 - 40 patients. The two planned treatments will be aerosolized furosemide and aerosolized saline, and will be given to each patient on two separate days. We failed to reach our enrollment goal, and ultimately enrolled 17 subjects for participation in Study 2b.

ELIGIBILITY:
Inclusion Criteria:

* Intractable dyspnea at rest or with minimal activity

Exclusion Criteria:

* Chronic congestive heart failure
* Liver or kidney disease
* Systemic lupus erythematosis (SLE)
* Receiving potassium supplementation or other indication of hypokalemia
* Major psychiatric disorders
* Furosemide hypersensitivity
* Not mentally competent and/or alert (unable to grant informed consent)
* Under 18 years old
* Not fluent in English
* Inadequate birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Banzett, PhD, Principal Investigator — Beth Israel Deaconess Hospital
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Banzett RB, Adams L, O'Donnell CR, Gilman SA, Lansing RW, Schwartzstein RM. Using laboratory models to test treatment: morphine reduces dyspnea and hypercapnic ventilatory response. Am J Respir Crit Care Med. 2011 Oct 15;184(8):920-7. doi: 10.1164/rccm.201101-0005OC. Epub 2011 Jul 21. PMID 21778294

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Aerosol Furosemide Study 2b Arm S: Inhalation of saline aerosol one one day then furosemide aerosol on another day. Baseline measurement 15 min; Inhalation over the course of 10-15 min.; outcome measurement 15 min. Watch for adverse effects 2 hours.
Period: Overall Study
Arm/Group | Aerosol Furosemide Study 2a | Aerosol Furosemide Study 2b Arm F | Experimental: Aerosol Furosemide Study 2b Arm S
Started | 7 | 9 | 8
Completed | 7 | 9 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Aerosol Furosemide Study 2b: Inhalation of furosemide aerosol or placebo saline aerosol over the course of 10-15 min. Single administration of furosemide aerosol on one treatment day, and a single administration of saline aerosol on a separate treatment day. Order of Furosemide Treatment Day and Placebo Treatment Day is randomized.
- Total: Total of all reporting groups
Arm/Group | Aerosol Furosemide Study 2a | Aerosol Furosemide Study 2b | Total
Number analyzed (Participants) | 7 | 17 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 8
  >=65 years | 4 | 12 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.14 (11.09) | 67.41 (11.41) | 67.92 (11.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 4 | 13 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 7 | 16 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 6 | 13 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 17 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Subject Rating of Breathing Discomfort (Dyspnea) Before and After Treatment.
Description: Subjects will rate breathing discomfort (dyspnea) during a 15 min exercise test using a visual analog scale before and after drug (or placebo) intervention. The treatment effect was measured as the rating of breathing discomfort rating before treatment minus the rating of breathing discomfort after treatment at equivalent work intensities.
  Outcome Measure Time Frame: subjects performed arm exercise to induce dyspnea for approximately 15 min before and after aerosol inhalation. the average number of minutes between end of drug administration and post-intervention breathing discomfort rating:
  Aerosol furosemide Study 2a arm: 38.7 minutes; Aerosol furosemide Study 2b arm: 21.8 minutes; Aerosol saline Study 2b arm: 21.3 minutes
Time Frame: 15 min
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Aerosol Furosemide Study 2b: Inhalation of furosemide aerosol. Baseline measurement 15 min; Inhalation over the course of 10-15 min.; outcome measurement 15 min. Watch for adverse effects 2 hours.
- Aerosol Saline Study 2b: Inhalation of saline aerosol . Baseline measurement 15 min; Inhalation over the course of 10-15 min.; outcome measurement 15 min. Watch for adverse effects 2 hours.
Arm/Group | Aerosol Furosemide Study 2a | Aerosol Furosemide Study 2b | Aerosol Saline Study 2b
Number analyzed (Participants) | 7 | 17 | 17
units on a scale | -1.86 (2.31) | -0.61 (1.61) | -0.15 (0.94)
Statistical Analysis 1: Comparison: Aerosol Furosemide Study 2b vs Aerosol Saline Study 2b; This is a paired t-test comparing the treatment effect of furosemide to the treatment effect of saline in each individual; Test type: Superiority; p = 0.35, t-test, 2 sided — The p-value is not adjusted for multiple comparisons and the a priori threshold for statistical significance was 0.05

2. Secondary Outcome: Urine Output - mL
Description: Diuresis is an expected effect of furosemide. To the extent that aerosol furosemide is absorbed in the blood, diuresis is an expected 'side effect' of this treatment.
  Following intervention, study team will measure urine output (mL). Study team will then rehydrate subject with an equal amount of liquid to their output.
Time Frame: Summation of total urine output (mL) at 1 hour following drug administration.
Population: The 17 participants in 'Aerosol furosemide Study 2b' and 'Aerosol saline Study 2b' are the results from the same 17 subjects on two different test days.
Measure: Mean (Standard Deviation); unit: ml of urine
Groups:
- Aerosol Furosemide Study 2b: Inhalation of furosemide aerosol over the course of 10-15 min.
  Across the study 2b, these subjects experienced a single administration of furosemide aerosol on one treatment day, and a single administration of saline aerosol on a separate treatment day. Order of Furosemide Treatment Day and Placebo Treatment Day is randomized.
- Aerosol Saline Study 2b: Inhalation of placebo saline aerosol over the course of 10-15 min.
  Across the study 2b, these subjects experienced a single administration of furosemide aerosol on one treatment day, and a single administration of saline aerosol on a separate treatment day. Order of Furosemide Treatment Day and Placebo Treatment Day is randomized.
Arm/Group | Aerosol Furosemide Study 2a | Aerosol Furosemide Study 2b | Aerosol Saline Study 2b
Number analyzed (Participants) | 7 | 17 | 17
ml of urine | 189.8 (236.2) | 573.6 (237.8) | 63.9 (93.9)
Statistical Analysis 1: Comparison: Aerosol Furosemide Study 2b vs Aerosol Saline Study 2b; Test type: Superiority; p < 0.001, t-test, 2 sided — The p-value is not adjusted for multiple comparisons, and the a priori threshold for significance was 0.05

ADVERSE EVENTS:
Groups:
- Aerosol Furosemide Study 2b: Inhalation of furosemide aerosol over the course of 10-15 min. Single administration of furosemide aerosol on one treatment day. Order of Furosemide Treatment Day and Placebo Treatment Day is randomized.
- Aerosol Saline Study 2b: Inhalation of placebo saline aerosol over the course of 10-15 min. Single administration of saline aerosol. Order of Furosemide Treatment Day and Placebo Treatment Day is randomized.
Arm/Group | Aerosol Furosemide Study 2a | Aerosol Furosemide Study 2b | Aerosol Saline Study 2b
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/7 | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No